CLINICAL TRIAL: NCT03529682
Title: The Effects of Circuit Training on Lower Extremities Functionality and Postural Control in Children With Cerebral Palsy
Brief Title: Circuit Training in Children With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Ünal Aras Değer, Senior Instructor, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/51-21
Record Dates: First submitted 2018-05-03; First posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Spastic Cerebral Palsy
Keywords: Circuit Exercise; Trunk Control; Functional Strength Training
MeSH Terms: conditions — Cerebral Palsy | interventions — Exercise; Circuit-Based Exercise; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Circuit Training Group (Experimental): Circuit exercise training will be given to the experimental group participants during 10 weeks, 60 minutes in a day and 3 times a week.
  Interventions: Other: exercise
- Control Group (Other): The control group participants will continue to their own previous physiotherapy approaches as the same as minimum 3 times a week and total 3 hours.
  Interventions: Other: control group

INTERVENTIONS:
Other: exercise — 10 minutes warm-up exercises and stretching exercises, 40 mınutes consecutive exercises (strengthening exercises for trunk and lower extremities) and 10 mınutes cooling down exercises and stretching exercises will be applied.
  Other Names: circuit training
  Arms: Circuit Training Group
Other: control group — 60 mınutes in a day and 3 times in a week traditional physiotherapy program will be applied
  Other Names: traditional physiotherapy
  Arms: Control Group

SUMMARY:
The aim of our study is to reveal the results of circuit training to be applied to the children with Cerebral Palsy (CP) for improving their muscular strength and trunk control and also to determine their effects in terms of activity limitations and participation limits.

DETAILED DESCRIPTION:
According the power analyzes totally 62 children, as 31 per each group, who were diagnosed with Spastic type CP and accepting participation for the study will be included in this study. For every case, socio demographic data and clinical features will be recorded. In the first session their gross motor function, muscular tonus in lower extremities, isometric strength of lower extremity muscles, functional muscular strength of the trunk and the lower extremities, walking speed and main mobility, functional motor performance will be assessed by a physiotherapist. Also satisfaction of children from the exercises, activity and participation level and quality of life will be evaluated. Then Covariant Focused Randomization Method will be used for having similarity in terms of factors such as; age, gender and motor function levels and also for having a balanced and equal case number of control and intervention group. The control group participants will continue to their own previous physiotherapy approaches (Bobath approach, traditional physiotherapy, etc.). "Circuit exercise training" will be given to the intervention group participants during 10 weeks, 3 times a week and that changes 50-60 minutes. At the end of the 10 weeks, the above evaluation parameters will be repeated

ELIGIBILITY:
Inclusion Criteria:

* The children who were diagnosed with Spastic type Cerebral Palsy.
* is aged between 6-18,
* is on the I,II and III levels according to Gross Motor Function Classification System

Exclusion Criteria:

* having any surgical operation related to lower extremities for the last 1 year,
* having botulinum toxin injection or intrathecal pump for the last 6 months,
* taking a new medicine or medicine change for the last 1 month,
* visual, hearing and epilepsy problem,
* inability to contınuously attend the exercise program,
* mental problem that could not be cooperated.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function will be evaluated | Change from baseline GMFS at 10 weeks
  As for the Gross Motor Function evaluation, the Gross Motor Function Scale (GMFS) will be used and only its D and E sections (standing, walking, running, jumping evaluation parts) will be used. By considering the instructions in to be tested parts in the scale, the case is expected to do the motor functions actively. Without the consideration of the quality of the movement, the case will be observed whether s/he started, was able to continue and completed the movement as well as whether s/he needed any support so that points between 0-3 will be given according to the level. The obtained total score determines the interaction severity of gross motor function

SECONDARY OUTCOMES:
Functional muscular strength of the trunk and the lower extremities will be evaluated. | Change from baseline Functional muscular strength at 10 weeks
  In order to determine the functional muscular strength of the body and the lower extremities, the step number will be recorded by taking straight step to the stair test and taking side step to the stair test in 15 seconds.
Isometric strength of bilateral lower extremity muscles and trunk muscles will be evaluated. | Change from baseline isometric strength at 10 weeks
  For the evaluation of isometric strength of bilateral lower extremity muscles and body muscles, a hand held dynamometer will be used which is in standard positions and independent from the gravity and the obtained measurement will be recorded by adjusting it to the body weight. The strength obtained by isometric contraction and by equipment resistance applied on key chosen muscles, will be recorded as a numerical value.
Muscular tonus in lower extremities will be evaluated. | Change from baseline muscular tonus at 10 weeks
  The muscular tonus in lower extremities will be evaluated as bilateral by Modified Ashworth Scale (MAS). The joint will be moved passively, fast and reverse to the muscular functions that will be tested in this scale -which is used for the determination of spasticity severity. According to the resistivity occurred, scoring is done between 0-4 points.
Walking speed and main mobility will be evaluated. | Change from baseline walking speed and main mobility at 10 weeks
  For the determination of walking speed and main mobility; timed up and go (TUG) test will be used. 3 meter walking distance will be recorded.
Functional motor performance will be evaluated. | Change from baseline functional motor performance at 10 weeks
  For the determination of functional motor performance; sitting and getting up test of Motor Assessment Scale will be used. Without a back and arm support, the chair sitting and getting up number in 1 minute will be recorded.
Satisfaction of children from the exercises will be evaluated. | At 10 weeks.
  For the measurement of satisfaction of children from the exercises to be applied, Physical Activity Enjoyment Scale (PACES) will be used. The children will be asked to mark the numbers suitable for themselves after reading child items in the 5 likert point scale. The points taken on the scale, change between 5 and 25.
Activity and participation level will be evaluated. | Change from baseline COPM at 10 weeks
  Canadian Occupational Performance Test (COPM) will be used in order to evaluate activity and participation level. COPM is an interview based method and the participant is asked to express the daily activities they needed, desired and they are not able to do. They are asked to express these activities under 3 headlines (self care activities, productivity and free time activities) and they are asked to determine these according to the priority for themselves. The first desire/problem is 10 points, and last is 1 point.
Quality of life will be evaluated. | Change from baseline LQSC at 10 weeks
  For the evaluation of life quality; Life Quality Scale for Children (LQSC) will be used (PedsQL) (5-7 age SP family reported model,5-7 age SP model, 8-12 age SP model, 13-18 age SP model). 23 questions will be used for the case which consists of 0-4 points and Working/Job Functions, Social, Physical and Emotional Functions in the last one month. The obtained point gives information about the life quality

CONTACTS AND LOCATIONS:
Overall Officials: UNAL DEGER, MSc, Principal Investigator — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus